CLINICAL TRIAL: NCT05685797
Title: Inflammatory Cytokine and Neuropeptide Study in Patients With Herpes Zoster
Brief Title: Biomarker Study in Patients With Herpes Zoster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-09-016
Record Dates: First submitted 2022-12-15; First posted 2023-01-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-07

CONDITIONS: Herper Zoster
Keywords: herpes zoster; cytokine; neurotransmitter
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- herpes zoster (acute) patients with intervention (Experimental): Patients with herpes zoster receiving 2 times of nerve block
  Interventions: Procedure: Herpes zoszter (acute)with inter vention
- patients with chronic herpes zoster receiving 2 times of nerve block (Experimental): Patients with herpes zoster receiving 2 times of nerve block
  Interventions: Procedure: Herpes zoszter (acute)with inter vention

INTERVENTIONS:
Procedure: Herpes zoszter (acute)with inter vention — nerve block

SUMMARY:
Investigators performed this study to investigate the expression levels inflammatory cytokine and neurotransmitters (calcitonin gene-related peptide (CGRP), substance P (SP), vasoactive intestinal peptide (VIP), and β-endorphin) in peripheral blood of participants with herpes zoster.

DETAILED DESCRIPTION:
Sudden and electrick shooting sensation of face is an important clinical feature of herpes zoster. The severe and excruciating nature of pain intensity associated with herpes zoster can impair the physical and psychosocial well-being of the patient, however, pathophysiologic mechanism of herpes zoster still remains unclear.

Recentrly, there have been a few studies suggesting biomarker levels in the blood and CSF level, however, further study is required to elucidate the action mechanism.

Up to 90% of patients can achieve pain reduction using medical therapy alone. However, 10% -15% of herpes zoster cases demonstrate a minimal response to medication with various side effects. Radiofrequency thermocoagulation (RFT) of the trigeminal ganglion is an alternative treatment option for patients who are poor candidates for microvascular decompression or show serious side effects to medication. Recent study revealed that RFT of the trigeminal ganglion resulted in Barrow Neurological Institute (BNI) pain scale I or II in 71.7% of patients, with a median time to recurrence of 36 months.

Although patients experience significant pain relief after RFT, it is uncertain whether inflammatory cytokine and neurocytokine (CGRP, substance P, VIP) are reduced.

ELIGIBILITY:
Inclusion Criteria:

* patients with NRS more than 4
* patients who failed medical treatment
* patients showing severe adverse reaction with medication

Exclusion Criteria:

* Patients showing allergic reaction to local anesthetics
* Patients with coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
serum level of inflammatory cytokine changes during 3 time period | Baseline, 1 week after tigeminal nerve block, 2 weeks after radiofrequency thermocoagulation
  inflammatory cytokine including Tumor necrosis factor-alpha, Interleukin-6 changes during 3 time period Higher score means worse outcome
serum level of neurotransmitter changes during 3 time period | Baseline, 1 week after tigeminal nerve block, 2 weeks after radiofrequency thermocoagulation
  neurotransmitter including Calcitonene gene related peptide, substance P, vasoactive intestitinal polypeptide changes during 3 time period Higher score means worse outcome

SECONDARY OUTCOMES:
Changes of numerical rating scale changes during 3 time period | Baseline, 1 week after tigeminal nerve block, 2 weeks after radiofrequency thermocoagulation
  numerical rating scale changes during 3 time period

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No